CLINICAL TRIAL: NCT00807235
Title: An Open Label, Multicenter, Phase 2, Pilot Evaluation of SURFAXIN®(Lucinactant) Delivered as an Aerosol Via Nasal Continuous Positive Airway Pressure (nCPAP) in the Prevention of Respiratory Distress Syndrome in Premature Infants
Brief Title: Feasibility Study of Aerosolized Surfaxin in the Prevention of Respiratory Distress Syndrome (RDS) in Premature Infants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Windtree Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KL4-CPAP-01
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Results first posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-05

CONDITIONS: Respiratory Distress Syndrome
Keywords: Lucinactant; Nasal continuous positive airway pressure (nCPAP); Respiratory distress syndrome (RDS); Pediatric; Premature
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen 1 (Experimental)
  Interventions: Drug: Aerosolized lucinactant
- Regimen 2 (Experimental)
  Interventions: Drug: Aerosolized lucinactant

INTERVENTIONS:
Drug: Aerosolized lucinactant — Aerosolized lucinactant via nCPAP over 3 hours. Up to 3 retreatments will be allowed over a 48 hour period with each retreatment separated by at least 3 hours.
  Other Names: KL₄Surfactant
  Arms: Regimen 1
Drug: Aerosolized lucinactant — Aerosolized lucinactant via nCPAP over 3 hours. Up to 3 retreatments will be allowed over a 48 hour period with each retreatment separated by at least 1 hour.
  Other Names: KL₄Surfactant
  Arms: Regimen 2

SUMMARY:
To evaluate the feasibility, safety and tolerability of aerosolized lucinactant delivered by nasal continuous positive airway pressure (nCPAP) for the prevention of respiratory distress syndrome (RDS) in premature infants.

DETAILED DESCRIPTION:
Use of a device in the early treatment of RDS that permits the effective aerosolization of an exogenous surfactant that also allows for the simultaneous delivery of continuous positive airway pressure would permit the delivery of surfactant to the distal airways without intubation. This approach could reduce the frequency of severity of the adverse events relative to endotracheal intubation and surfactant administration via bolus.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 28-32 completed weeks, inclusive
* Placement of arterial line
* Successful initiation of nCPAP
* Informed Consent

Exclusion Criteria:

* Heart rate that cannot be stabilized >100 bpm within 5 minutes of birth
* Five (5) minute Apgar score ≤ 3
* Major congenital malformation(s) diagnosed antenatally or noted immediately after birth
* Other disease(s) or conditions potentially interfering with cardiopulmonary function
* Mother with prolonged rupture of membranes > 2 weeks
* Known or suspected chromosomal abnormality
* Need for chest compressions or administration of epinephrine, bicarbonate, or fluid boluses in the delivery room
* Need for mechanical ventilation within 30 minutes of birth

Ages: 15 Minutes to 30 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2005-01; Primary Completion 2005-08 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Finer, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Medical Center - Hillcrest, San Diego, California, United States

REFERENCES:
- [Result] Finer NN, Merritt TA, Bernstein G, Job L, Mazela J, Segal R. An open label, pilot study of Aerosurf(R) combined with nCPAP to prevent RDS in preterm neonates. J Aerosol Med Pulm Drug Deliv. 2010 Oct;23(5):303-9. doi: 10.1089/jamp.2009.0758. PMID 20455772

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Neonates were enrolled between January and August, 2005. This was an open-label study with 2 treatment groups (Regimen 1 and Regimen 2). Eligible neonates were sequentially enrolled and stratified by GA into 2 strata for each regimen. For each regimen, enrollment in Stratum 1 (30 to 32 GA) was completed before enrollment in Stratum 2 (28 to 29 GA).
Groups:
- Lucinactant - 3 Hour Interval: Aerosolized Lucinactant via nasal continuous positive airway pressure (nCPAP) w/ Retreatment after 3 hours
- Lucinactant - 1 Hour Interval: Aerosolized Lucinactant via nasal continuous positive airway pressure (nCPAP) w/ Retreatment after 1 hour
Period: Overall Study
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Started | 11 | 6
Completed | 10 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 6 | 17
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 11 | 6 | 17
Gestational Age [Mean (Standard Deviation); unit: weeks] | 29.8 (1.40) | 30.7 (0.99) | 30.1 (1.31)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Respiratory Distress Syndrome
Time Frame: 24 hours
Population: This was a phase 2, pilot, estimation study. Hence, sample size calculations were not performed.
  All enrolled infants analyzed (intent-to-treat).
Measure: Number; unit: participants
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
participants | 4 | 0

2. Secondary Outcome: Area Under the Curve (AUC) for Fraction of Inspired Oxygen (FiO₂)
Description: AUC for FiO₂calculated using the trapezoidal rule. Missing data imputed using last observation carried forward
Time Frame: 0.5, 1, 2, 4, 6, 12, 18, 24, 36, 48, 60, 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent O₂*hours
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
percent O₂*hours | 0.36 (0.15) | 0.25 (0.08)

3. Secondary Outcome: Arterial Alveolar (a/A) O₂Ratio
Description: a/A ratio is a relative way to judge the lungs ability to transport O₂. It compares the partial pressure of O₂in the alveoli (A) to the partial pressure of O₂in the artery (a). It is calculated by dividing the partial pressure of O₂in the artery, abbreviated PaO2, by the partial pressure of O₂in the alveoli using the alveolar gas equation, abbreviated PAO2. A value of 0.80 or above is normal, a value of 0.60 or below may be incompatible with spontaneous breathing, and a value below 0.22 indicates severe lung disease.
Time Frame: 72 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg over mm Hg (ratio of pressures)
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
mm Hg over mm Hg (ratio of pressures) | 0.46 (0.25) | 0.53 (0.29)

4. Secondary Outcome: Time to Meet Failure Criteria
Description: Failure criteria defined as rescue with bolus surfactant and mechanical ventilation
Time Frame: Through 28 days
Population: This was a phase 2, pilot, estimation study. Hence, sample size calculations were not performed.
  All enrolled infants analyzed (intent-to-treat). Time in days calculated for neonates who met failure criteria (3 for Regimen 1, 2 for Regimen 2)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
days | 0.49 (0.38) | 0.30 (0.35)

5. Secondary Outcome: Number of Participants With Bronchopulmonary Dysplasia (BPD)
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
participants | 1 | 1

6. Secondary Outcome: Number of Participants Alive and Without BPD
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
participants | 10 | 5

7. Secondary Outcome: Number of Participants With Intraventricular Hemorrhage (IVH)/Periventricular Leukomalacia (PVL)
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
participants | 1 | 0

8. Secondary Outcome: Number of Participants With Patent Ductus Arteriosus (PDA)
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
participants | 3 | 3

9. Secondary Outcome: Number of Participants With Necrotizing Enterocolitis (NEC)
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
participants | 0 | 0

10. Secondary Outcome: Number of Participants With Pulmonary Hemorrhage
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
participants | 0 | 0

11. Secondary Outcome: Number of Participants With Acquired Sepsis
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
participants | 2 | 1

12. Secondary Outcome: Incidence of Mortality
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
participants | 0 | 0

13. Secondary Outcome: Number of Participants With Air Leak
Time Frame: 28 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Number analyzed (Participants) | 11 | 6
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Lucinactant - 3 Hour Interval | Lucinactant - 1 Hour Interval
Serious Adverse Events (participants affected / at risk) | 5/11 | 1/6
Other Adverse Events (participants affected / at risk) | 11/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lucinactant - 3 Hour Interval (N=11) | Lucinactant - 1 Hour Interval (N=6)
Sepsis neonatal (Infections and infestations) | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Neonatal apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension NOS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lucinactant - 3 Hour Interval (N=11) | Lucinactant - 1 Hour Interval (N=6)
Anaemia neonatal (Blood and lymphatic system disorders) | 2 | 3
Bradycardia NOS (Cardiac disorders) | 1 | 3
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 4 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Oedema NOS (General disorders) | 1 | 1
Jaundice neonatal (Hepatobiliary disorders) | 3 | 1
Abscess NOS (Infections and infestations) | 1 | 0
Pneumonia NOS (Infections and infestations) | 0 | 1
Sepsis neonatal (Infections and infestations) | 2 | 1
Oxygen saturation decreased (Investigations) | 6 | 3
Acidosis NOS (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 2
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis NOS (Metabolism and nutrition disorders) | 3 | 0
Feeding problem in newborn (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Agitation neonatal (Psychiatric disorders) | 1 | 0
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal passage irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Neonatal apnoeic attach (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Intraventricular haemorrhage neonatal (Vascular disorders) | 1 | 0
Neonatal hypotension (Vascular disorders) | 1 | 0
Pulmonary hypertension NOS (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days